CLINICAL TRIAL: NCT02959060
Title: An Open-Label, Single-Sequence Study to Evaluate the Effect of Rifampin on the Single-dose Pharmacokinetics of BMS-986177 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Rifampin on the Single-dose Pharmacokinetics of BMS-986177 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CV010-014
Record Dates: First submitted 2016-11-07; First posted 2016-11-08 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-986177 and Rifampin (Experimental)
  Interventions: Drug: BMS-986177; Drug: Rifampin

INTERVENTIONS:
Drug: BMS-986177 — Single dose of BMS-986177 and multiple doses of Rifampin
Drug: Rifampin — Single dose of BMS-986177 and multiple doses of Rifampin

SUMMARY:
This study is to evaluate the effect of rifampin on the single-dose pharmacokinetics (PK) of BMS-986177 in healthy participants with parameters like Cmax, AUC(INF), AUC(0-T)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Healthy men and women (not of child bearing potential) as determined by medical history, surgical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests including coagulation parameters.
3. Subjects with body mass index of 18 to 30 kg/m2, inclusive and with normal kidney function.
4. Women participants must have documented proof that they are not of childbearing potential.
5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with BMS-986177 plus 5 half-lives (3 days) plus 90 days (duration of sperm turnover) for a total of 93 days after completion of BMS-986177 treatment.

Exclusion Criteria:

1. Any significant acute or chronic medical illness, including any other condition listed as a contraindication in the rifampin package insert
2. History of recurrent headaches, dizziness, chronic diarrhea, gastroesophageal reflux disease, dyspepsia, gastrointestinal ulcer disease, recurrent urinary tract infections, hypermenorrhea and recurrent candida infections, abnormal bleeding, history of hemophilia, Rosenthal syndrome, FXIa deficiency, or other coagulopathies.
3. Recent surgery, head injury, blood transfusion, systemic lupus erythamatous, aneurysm, drug or alcohol abuse and use of tobacco or nicotine containing products in past six months.
4. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs, or clinical laboratory determinations beyond what is consistent with the target population
5. History of allergy to BMS-986177, FXIa inhibitors , rifampin or related compounds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Days1-15
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Days1-15
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Days1-15

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and death | Screening- until 30 days after discontinuation of dosing or subject's participation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Perera V, Wang Z, Lubin S, Christopher LJ, Chen W, Xu S, Seiffert D, DeSouza M, Murthy B. Effects of rifampin on the pharmacokinetics and pharmacodynamics of milvexian, a potent, selective, oral small molecule factor XIa inhibitor. Sci Rep. 2022 Dec 23;12(1):22239. doi: 10.1038/s41598-022-25936-2. PMID 36564395
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx